CLINICAL TRIAL: NCT00148590
Title: Memantine add-on to Risperidon for Treatment of Negative Symptoms and Cognitive Dysfunction in Patients With Acute Schizophrenia: Results of a Proof of Concept Study
Brief Title: Memantine for the Prevention of Cognitive Dysfunction and Negative Symptoms in Patients With Acute Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: M. Schaefer, MD (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, M. Schaefer, MD, Professor of Psychiatry, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MIND 1; 02T-247 (SMRI)
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia
Keywords: Memantine; Negative syndrome; Schizophrenia; Cognitive impairment; Glutamate
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine plus Risperidone (Active Comparator): 6 weeks 20 mg Memantine as add-on treatment to Risperidone
  Interventions: Drug: Memantine
- Placebo plus Risperidone (Placebo Comparator): 6 weeks 20 mg Placebo as add-on treatment to Risperidone
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Daily dose of 20 mg Memantine add-on to Risperidone vs Placebo add-on to Risperidone
  Other Names: Akatinol
  Arms: Memantine plus Risperidone
Drug: Placebo — Daily dose of 20 mg Memantine add-on to Risperidone vs Placebo add-on to Risperidone
  Arms: Placebo plus Risperidone

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a 6 weeks memantine add-on to risperidon treatment for the prevention of cognitive dysfunction and negative symptomatology in patients with acute schizophrenia.

Psychopathological changes were assessed with the Positive and Negative Syndrome Scale (PANSS) at baseline and after 2, 4, 6, 12, and 24 weeks. Cognitive function were measured at baseline and week 6, and 24 by the California Verbal Learning Test, Benton Learning Test, Digit Span Forward and Backward Test, Continuous Performance Test, Stroop Test, Trail-Making Test, Verbal Fluency Test, and Wisconsin Card Sorting Test.

DETAILED DESCRIPTION:
This study examines the efficacy and safety of a 6 weeks memantine add-on to risperidon treatment for the prevention of cognitive dysfunction and negative symptomatology in patients with acute schizophrenia. The trail is double-blind, prospective, randomized, placebo-controlled, parallel-group and consisting of a 'placebo-run-in' period, treatment, and follow-up periods. Study personnel and participants were blinded to group assignment. In the 'run-in' period, patients received Lorazepam for the treatment of anxiety and tension states for two weeks before starting antipsychotic therapy. After the 'run-in' period treatment, patients began receiving antipsychotic therapy with Risperidon with continuous concomitant administration of Memantine, 20 mg/d, or placebo for six weeks. Adherence was assessed at each clinic visit by pill count. In cases of anxiety and tension states, an experienced psychiatrist decided whether patients should receive Lorazepam, 5 mg/d, as rescue medication in addition to the study medication (Memantine or placebo), to which the patients remained blinded. In cases of pseudo parkinsonism patients were allowed to receive Biperiden, up to 8 mg/d, and for the treatment of patients suffering from sleep disorders Zopiclon (15 mg/d) was allowed. The consumption of alcohol and drugs were not allowed during the trial. In both study parts, psychiatric assessments were performed at baseline as well as after 2; 4; 6; 12 and 24 weeks after treatment (that is, during the follow-up period). The neuropsychological examination was performed at baseline, and after 6 and 24 weeks. Psychiatric changes, adverse events, laboratory values, dose adjustments of the antipsychotic therapy, and possible pharmacologic adverse effects were systematically monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (DSM-IV)
* Age 18 to 40
* Exacerbation of an acute schizophrenic episode (PANSS positive score > 20)
* At least one previous schizophrenic episode
* Informed consent
* Subjects must be considered by the investigator to be compliant
* Subjects must have an educational level and a degree of understanding such that they can meaningfully communicate with the investigator

Exclusion Criteria:

* Axis I disorder other than schizophrenia within 12 months, e.g. schizoaffective disorder
* Severe negative symptomatology (PANNS negative score >20 points)
* Duration of schizophrenia > 5 years
* Dependency on alcohol or addictive drugs within 6 months of the baseline evaluation
* Contraindication of risperidone
* Significant neurological, cardiovascular, hepatic, renal, metabolic, or other medical diseases or any clinically relevant abnormalities in laboratory tests
* Prior ECT-treatment, metal implantations
* Female subjects during pregnancy and breastfeeding
* Female subjects within childbearing years who were not using adequate birth control
* Patients who are judged by the investigator to be at serious suicide risk

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Changes in PANSS negative subscore between memantine and placebo treatment | during trial

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schaefer, MD, Principal Investigator — Charite Campus Mitte; Dept. of Psychiatry and Psychotherapy and Department of Psychiatry, Kliniken Essen-Mitte, Essen
Locations (1):
- Charité Universitaetsmedizin Berlin; Campus Charité Mitte; Dept. for Psychiatry and Psychotherapy, Berlin, Germany

REFERENCES:
- [Derived] Schaefer M, Sarkar S, Theophil I, Leopold K, Heinz A, Gallinat J. Acute and Long-term Memantine Add-on Treatment to Risperidone Improves Cognitive Dysfunction in Patients with Acute and Chronic Schizophrenia. Pharmacopsychiatry. 2020 Jan;53(1):21-29. doi: 10.1055/a-0970-9310. Epub 2019 Aug 7. PMID 31390660